CLINICAL TRIAL: NCT02464098
Title: Epidemiology of Diarrheal Diseases in Pediatric Oncology Patients
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EPIGUT
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Diarrhea
Keywords: Hematological Malignancies; Solid Tumors; Hematopoietic Stem Cell Transplantation (HSCT); Childhood Cancer; Polymerase Chain Reaction (PCR)
MeSH Terms: conditions — Diarrhea; Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All stool, blood and respiratory samples will be saved frozen for future testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Participants with diagnosis of hematological malignancy or solid tumor.
- Group 2: Participants undergoing hematopoietic stem cell transplantation (HSCT).

SUMMARY:
Diarrhea is a common problem in the pediatric population. Children with cancer are especially at increased risk for gastrointestinal infection-related morbidity and mortality due to their ongoing immunosuppression. However, the epidemiology of diarrheal illnesses in immunocompromised children is poorly understood. In the past, many or most cases of gastroenteritis have gone undiagnosed, largely due to a lack of sensitive diagnostic tests and a presumption that a large proportion of cases are due to treatment, rather than infections. The availability of new diagnostic tests that detect many gastrointestinal pathogens simultaneously offers the first opportunity to gain a comprehensive picture of the causes of infectious diarrhea in children with cancer.

Researchers at St. Jude Children's Research Hospital want to learn about the epidemiology of diarrheal diseases in pediatric oncology patients utilizing broadly multiplexed, automated PCR.

DETAILED DESCRIPTION:
This study plans to enroll participants in two groups:

* GROUP 1: Participants with hematologic malignancies or solid tumors.

  * Participants who agree to take part in this research study will have stool samples collected at diagnosis (baseline sample) and each month thereafter for 12 months from the time of enrollment. Stool samples will be screened for different types of microbes that may be present. For participants who develop diarrhea during these 12 months, three additional stool samples will be collected on Day 0, Day 7 and Day 14; two blood samples and mid-turbinate nasal swab will be collected as well on Day 0 and Day 7 of the first observed diarrheal episode to screen for additional microbes that may be the cause of the diarrhea.
* GROUP 2: Participants who are hematopoietic stem cell transplant (HSCT) patients.

  * Participants who agree to take part in this research study will have stool samples collected within one week prior to conditional chemotherapy (baseline sample) and weekly thereafter for a total of 16 weeks (pre- and early post-engraftment periods), followed by monthly for 8 months. Stool samples will be screened for different types of microbes that may be present. For participants who develop diarrhea, three additional stool samples will be collected on Day 0, Day 7 and Day 14; two blood samples and mid-turbinate nasal swab will be collected as well on Day 0 and Day 7 of the first observed diarrheal episode to screen for additional microbes that may be the cause of the diarrhea. For GROUP 2 participants, two diarrheal episodes will be studied per patient: the first diarrheal episode during the pre-engraftment period, and the first diarrheal episode during the post-engraftment period.

Participants with a change in cancer treatment plan enrolled on study: Group 1 participants who experience a change in their cancer treatment plan necessitating an allogeneic stem cell transplant will be taken off study for group 1 and offered the opportunity to consent to group 2 Participants who chooses to then enroll on group 2 will complete the 12-month study requirements as defined in the protocol for group 2 participants.

General health information from participant medical records and other health-related information about symptoms will also be obtained at the time of collection of the samples.

PRIMARY OBJECTIVE:

* To assess the prevalence of microbial pathogens in the stool of pediatric oncology patients with diarrheal illness.

SECONDARY OBJECTIVES:

* To describe the clinical course, symptomatology, morbidity and mortality associated with diarrheal diseases in pediatric oncology patients at St. Jude Children's Research Hospital.
* Evaluate the performance of the multiplex polymerase chain reaction (PCR) assay for the diagnosis of infectious diarrhea in comparison to the standard of care methods.

ELIGIBILITY:
Inclusion Criteria:

* Equal to or less than 18 years of age.
* GROUP 1: Patients diagnosed in the preceding 14 days with confirmed diagnosis at St. Jude of a new hematological malignancy or solid tumor in the preceding 14 days, OR patients diagnosed with a new hematological malignancy or solid tumor and has initiated chemotherapy within the previous 72 hours from enrollment.
* GROUP 2: Patients scheduled to receive conditioning for hematopoietic stem cell transplant (HSCT) in the subsequent 7 days.
* Parent or legal guardian willing and able to give informed consent and comply with study requirements.
* Anticipated to be available for all study visits.

Exclusion Criteria:

* Patients from GROUP 1 (diagnosed in the preceding 14 days with a new hematological malignancy or solid tumor) who underwent HSCT in the previous 12 months.
* Has any condition that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be pediatric oncology patients including patients with recent diagnoses of solid tumor or hematologic malignancy, or patients undergoing hematopoietic stem cell transplant.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency by pathogen type of infectious pathogens | at 12 months
  Descriptive statistics of infectious pathogens identified in diarrheal stools from PCR testing will be summarized.
Proportion by pathogen type of infectious pathogens | at 12 months
  Descriptive statistics of infectious pathogens identified in diarrheal stools from PCR testing will be summarized.

SECONDARY OUTCOMES:
Frequency of symptoms | at 12 months
  Descriptive statistics of symptoms, clinical course, morbidity and mortality in patients with diarrhea will be summarized.
Proportion of symptoms | at 12 months
  Descriptive statistics of symptoms, clinical course, morbidity and mortality in patients with diarrhea will be summarized.
Number of infectious pathogens identified by multiplex PCR assay versus standard tests | at 12 months
  Infectious pathogens of diarrheal stools identified by the multiplex PCR assay will be compared descriptively against those identified by standard testing, and McNemar's test will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Randall T. Hayden, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols